CLINICAL TRIAL: NCT03015467
Title: Alteration of Intestinal Microflora and Efficacy and Safety of Fecal Microbiota Transplantation for Severe Acute Pancreatitis
Brief Title: Fecal Microbiota Transplantation (FMT) for Severe Acute Pancreatitis(SAP)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AM-FMT-SAP
Record Dates: First submitted 2017-01-03; First posted 2017-01-10 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Acute Pancreatitis; Intestinal Bacteria Flora Disturbance; Intestinal Dysfunction; Fecal Microbiota Transplantation
Keywords: acute pancreatitis; intestinal mucosal barrier; Fecal Microbiota Transplantation
MeSH Terms: conditions — Pancreatitis | interventions — Fecal Microbiota Transplantation; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment for part 1 (Active Comparator): Fecal Microbiota Transplantation (FMT) and traditional treatments according to associated guidelines will be used in patients with severe acute pancreatitis(SAP) in part 1.
  Interventions: Other: Fecal Microbiota Transplantation
- Placebo for part 2 (Placebo Comparator): The traditional treatments and normal saline (NS) according to associated guidelines will be used in patients with severe acute pancreatitis(SAP) in part 2.
  Interventions: Other: normal saline

INTERVENTIONS:
Other: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation and the traditional treatments for Acute Pancreatitis with gut mucosal barrier dysfunction and unbalance of gut microflora in part 1
  Other Names: Fecal Microbiota Transplantation (FMT)
  Arms: treatment for part 1
Other: normal saline — normal saline and the traditional treatments for Acute Pancreatitis with gut mucosal barrier dysfunction and unbalance of gut microflora in part 2
  Other Names: normal saline (NS)
  Arms: Placebo for part 2

SUMMARY:
Severe acute pancreatitis is an acute and rapid progress of the digestive system disease.Most patients with severe pancreatitis associated with intestinal mucosal barrier dysfunction.Intestinal microflora,an important part of the intestinal mucosal barrier, play an important role in the development process in the course of severe acute pancreatitis. At this stage of the study that infection of pancreas and other organs is the leading cause of death in patients with severe acute pancreatitis，and the main pathogens from intestinal micro-organisms， but the intestinal flora changes did not be mentioned. Fecal Microbiota Transplantation that has been used for treatment of inflammatory bowel disease and Clostridium difficile infection may be a new technology for regulation of intestinal mucosal dysfunction and intestinal flora unbalance.

DETAILED DESCRIPTION:
Patients with acute pancreatitis will be assessed depending on APACHE II and CT score and all of them also will be separated into two parts depending on acceptation or refusal of FMT. Blood specimens from patients will be collected to analysis inflammatory factors，and fecal microbiota samples will be detection.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of acute pancreatitis: elevated serum amylase and/or lipase levels (more than 3-fold the upper reference limit) and evidence of pancreatitis on computed tomography (CT) of the abdomen;
2. No chronic diseases of the digestive system ;
3. No chronic diseases of the urinary system;
4. No chronic metabolic disease;
5. No chronic disease of immune system
6. No chronic disease of mental disease
7. no acute intestinal disease; taking antibiotics anti-inflammatory drugs and history of probiotics for one month;
8. No use of addictive drugs and immune inhibitors

Exclusion Criteria:

1. not to match the standard of AP
2. with chronic diseases of the digestive system;
3. with chronic diseases of the urinary system;
4. with chronic metabolic disease;
5. with chronic disease of immune system
6. with chronic disease of mental disease
7. with acute intestinal disease; taking antibiotics anti-inflammatory drugs and history of probiotics for one month;pregnancy and lactation women
8. with use of addictive drugs and immune inhibitors
9. exceed the age limits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Mortality | 3 months

SECONDARY OUTCOMES:
C-reactive protein（CRP） | 2-4 weeks
Diamine oxidase（DAO） | 2-4 weeks
Interleukin | 2-4 weeks
tumor necrosis factor-a(TNF-a) | 2-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Li Fang, Ph.D, Study Chair — First Affiliated Hospital of Chengdu Medical College
Locations (1):
- IEC of Chengdu Medical College, Chendu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noor MT, Radhakrishna Y, Kochhar R, Ray P, Wig JD, Sinha SK, Singh K. Bacteriology of infection in severe acute pancreatitis. JOP. 2011 Jan 5;12(1):19-25. PMID 21206096
- [Background] Murphy SF, Rhee L, Grimm WA, Weber CR, Messer JS, Lodolce JP, Chang JE, Bartulis SJ, Nero T, Kukla RA, MacDougall G, Binghay C, Kolodziej LE, Boone DL. Intestinal epithelial expression of TNFAIP3 results in microbial invasion of the inner mucus layer and induces colitis in IL-10-deficient mice. Am J Physiol Gastrointest Liver Physiol. 2014 Nov 1;307(9):G871-82. doi: 10.1152/ajpgi.00020.2014. Epub 2014 Sep 18. PMID 25234043
- [Background] Wu LM, Sankaran SJ, Plank LD, Windsor JA, Petrov MS. Meta-analysis of gut barrier dysfunction in patients with acute pancreatitis. Br J Surg. 2014 Dec;101(13):1644-56. doi: 10.1002/bjs.9665. Epub 2014 Oct 21. PMID 25334028
- [Background] Fishman JE, Levy G, Alli V, Zheng X, Mole DJ, Deitch EA. The intestinal mucus layer is a critical component of the gut barrier that is damaged during acute pancreatitis. Shock. 2014 Sep;42(3):264-70. doi: 10.1097/SHK.0000000000000209. PMID 24978882
- [Background] Schwender BJ, Gordon SR, Gardner TB. Risk factors for the development of intra-abdominal fungal infections in acute pancreatitis. Pancreas. 2015 Jul;44(5):805-7. doi: 10.1097/MPA.0000000000000334. PMID 25872170
- [Background] Hall JC, Crawford HC. The conspiracy of autophagy, stress and inflammation in acute pancreatitis. Curr Opin Gastroenterol. 2014 Sep;30(5):495-9. doi: 10.1097/MOG.0000000000000097. PMID 25003605
- [Background] Senocak R, Yigit T, Kilbas Z, Coskun AK, Harlak A, Mentes MO, Kilic A, Gunal A, Kozak O. The Effects of Total Colectomy on Bacterial Translocation in a Model of Acute Pancreatitis. Indian J Surg. 2015 Dec;77(Suppl 2):412-8. doi: 10.1007/s12262-013-0855-y. Epub 2013 Jan 31. PMID 26730036
- [Background] Bongaerts GP, Severijnen RS. A reassessment of the PROPATRIA study and its implications for probiotic therapy. Nat Biotechnol. 2016 Jan;34(1):55-63. doi: 10.1038/nbt.3436. PMID 26744983
- [Background] Hansson GC, Johansson ME. The inner of the two Muc2 mucin-dependent mucus layers in colon is devoid of bacteria. Gut Microbes. 2010 Jan;1(1):51-54. doi: 10.4161/gmic.1.1.10470. PMID 21327117
- [Background] Zhang XP, Zhang J, Song QL, Chen HQ. Mechanism of acute pancreatitis complicated with injury of intestinal mucosa barrier. J Zhejiang Univ Sci B. 2007 Dec;8(12):888-95. doi: 10.1631/jzus.2007.B0888. PMID 18257123